CLINICAL TRIAL: NCT04330768
Title: Platelet Rich Fibrin(PRF) Versus Pulp Capping in Treatment of Dental Pulp Exposure:Randomized Clinical Trial
Brief Title: Platelet Rich Fibrin(PRF) Injection for Treatment of Dental Pulp Exposure:Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina mounir elkady, Lecturer at conservative department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0555
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Dental Pulp Exposure; Dental Caries
MeSH Terms: conditions — Dental Pulp Exposure; Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF (Experimental)
  Interventions: Procedure: PRF pulp capping
- MTA (Active Comparator)
  Interventions: Procedure: MTA pulp capping

INTERVENTIONS:
Procedure: PRF pulp capping — PRF is injected in the site of exposure
  Arms: PRF
Procedure: MTA pulp capping — conventional pulp capping procedure
  Arms: MTA

SUMMARY:
platelet rich fibrin(PRF) obtained from patient from patient blood sample (before start of treatment)is injected in the site of exposure of exposure(intervention group) control group will receive normal pulp capping procedure by MTA follow up will be one year

DETAILED DESCRIPTION:
intervention group:patient with deep caries lesion ,free from sign and symptoms of irreversible pulpitis the blood sample will be taken before the beginning of dental treatment..PRF will be obtained by blood centrifugal and injected in the site of exposure covered by glass ionomer restoration control group: patient with same condition will receive pulp capping procedure by MTA followed by glass ionomer restoration

ELIGIBILITY:
Inclusion Criteria:

* deep carious lesion- no sign of irreversible pulpitis

Exclusion Criteria:

* old age- periapical lesion-

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
pulp vitality | After 1 year
  no sign of irreversible pulpitis or pulpal necrosis

IPD SHARING:
Plan to Share IPD: No